CLINICAL TRIAL: NCT00616564
Title: Multicenter Phase II Trial of High-Dose Interleukin (IL-2) With Priming and Concomitant Sargramostim (GM-CSF) in Patients With Advanced Melanoma
Brief Title: Phase II Trial of (IL-2) With Priming and (GM-CSF) in Patients With Advanced Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mt. Sinai Medical Center, Miami (Other)
Collaborators: Bayer (Industry); Chiron Corporation (Industry)
Responsible Party: Principal Investigator, Jose Lutzky, Principal Investigator Jose Lutzky, M.D., Mt. Sinai Medical Center, Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEL0105
Record Dates: First submitted 2008-02-04; First posted 2008-02-15 (Estimated); Last update posted 2012-05-03 (Estimated); Status verified 2012-05

CONDITIONS: Malignant Melanoma
Keywords: GM-CSF; Interleukin; IL-2; Sargrostim
MeSH Terms: conditions — Melanoma | interventions — Granulocyte-Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: GM-CSF — Concomitant Priming with GM-CSF

SUMMARY:
High-dose IL-2 treatment for metastatic melanoma has been approved by the FDA in 1998. Studies of GM-CSF plus IL-2 have not addressed the approved dose and schedule. This protocol will study the combination of HD-IL2 and GM-CSF given the potential synergistic interactions discussed above.

DETAILED DESCRIPTION:
The primary objectives of this phase II multicenter trial are to:

Determine the 1 and 2-year survival of patients treated according to protocol. Assess the safety and toxicity of this regimen in this patient population.

The secondary objectives are to:

Determine the freedom from progression (FFP). Measure the response rate (RR). Obtain immunological data from the use of this regimen in vivo (as separate project: Moffitt?).

The proposed study is a multicenter phase II trial of HD-IL-2 in combination with GM-CSF. GM-CSF will be started 7 days before day 1 of HD-IL-2 and will be continued for 4 weeks to day 28, encompassing two cycles of HD-IL2. The first 9 patients will be closely monitored for unexpected toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of melanoma with measurable disease
* Patients with stage IV or unresectable advanced melanoma
* Age at least 16 years.
* ECOG performance status of 0-1
* Life expectancy > 3 months
* Adequate major organ function to tolerate therapy, as defined by:

  * Total bilirubin 2.0 mg/dL.
  * Creatinine 1.8 mg/dL.
  * WBC 3,000/mm3.
  * Platelet count 100,000/mm3.
* Patients 50 years of age with one or more cardiac risk factors must demonstrate normal exercise stress test, stress thallium test, or comparable cardiac ischemia evaluation
* Left ventricular ejection fraction > 40%
* Women of childbearing age must agree to use barrier method birth control and demonstrate a negative pregnancy test prior to initiation of protocol therapy. Periodic negative urine pregnancy tests will also be required.
* Patients must give written informed consent

Exclusion Criteria:

* No prior HD- IL-2 for stage IV/unresectable advanced disease. Prior low dose IL-2 is allowed.
* No more than 2 prior chemotherapy regimens are allowed.
* No active CNS metastases. Treated CNS metastases without recurrence or progression for > 8 weeks are allowed.
* No concurrent use of systemic corticosteroids
* Pregnant and/or lactating are excluded
* No concurrent antineoplastic treatments, including chemotherapy, biologic response modifiers, radiation, vaccines, or other experimental therapies.
* No treatment for melanoma within the previous 4 weeks.

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2006-02; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Primary Objective | one - two years
  Determine the 1 and 2-year survival of patients treated according to protocol. Assess the safety and toxicity of this regimen in this patient population

CONTACTS AND LOCATIONS:
Overall Officials: Jose Lutzky, M.D., Study Chair — Mount Sinai Medical Center Miami Beach
Locations (2):
- United States (2):
  - Jose Lutzky, MD, Miami Beach, Florida
  - David Lawson, MD, Atlanta, Georgia